CLINICAL TRIAL: NCT01876381
Title: A Phase 2, Multi-center, Open-label, Dose-finding Trial to Investigate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of OPC-41061 in Patients With Chronic Renal Failure Undergoing Hemodialysis or Hemodiafiltration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-12-007; JapicCTI-132147 (Other: JAPIC)
Record Dates: First submitted 2013-06-09; First posted 2013-06-12 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2017-11

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-41061 (Experimental)
  Interventions: Drug: OPC-41061

INTERVENTIONS:
Drug: OPC-41061 — The maximum number of days of administration will be 8 days (8 doses) in total 4 days each in the dose-escalation period and intermittant administration period. The investigational medicinal product (IMP) will be administered once daily after breakfast

SUMMARY:
To investigate the safety, pharmacokinetics, pharmacodynamics, and efficacy of OPC-41061 in patients with chronic renal failure undergoing hemodialysis or hemodiafiltration using variables, such as daily urine volume and increase in interval body weights between hemodialysis or hemodiafiltration, in 4-day intermittant administration (excluding the days of hemodialysis or hemodiafiltration) at the dose fixed during the dose-escalation period

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic renal failure who are undergoing hemodialysis or hemodiafiltration three times a week
* Subjects between the ages of 20 and 80, inclusive (at time of informed consent)
* Subjects who are inpatients or who can be admitted to the trial site for the duration of the trial period
* Subjects who, together with their partner, are able to practice one of the specified contraceptive methods until 4 weeks after the final trial drug administration
* Patients who are capable of providing written informed consent themselves before any trial-related procedures are performed

Exclusion Criteria:

* Subjects with a complication of urinary impairment due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
* Subject with daily urine volume less than 500 mL
* Subject with Cardiac function of NYHA class 4
* Subjects with serious ischemic heart disease, who are judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial
* Subjects with serious arrhythmia, who are judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial
* Subjects who are concomitantly undergoing peritoneal dialysis
* Subjects with ascites due to cirrhosis or cancer, requring medical treatments
* Subjects with any of the following medical histories:

  * History of cerebrovascular disorder or coronary artery disease within 4 weeks prior to informed consent
  * History of hypersensitivity or idiosyncratic reaction to benzazepine derivatives such as mozavaptan hydrochloride or benazepril hydrochloride
* Subjects with any of the following abnormal laboratory values:

  * Hemoglobin lower than 8.0 g/dL, total bilirubin higher than 3.0 mg/dL, ALT (GPT) or AST (GOT) 2 times the upper limit of the reference range of the trial site, serum sodium higher than the upper limit of the reference range of the trial site, serum sodium lower than 125mEq/L
* Subjects with serum potassium higher than 6.0mEq/L and abnormal findings inappropriate for inclusion in the trial are observed by 12-lead ECG
* Subjects who are unable to sense thirst or who have difficulty with fluid or food intake
* Subjects who have participated in any other clinical trial or post-marketing clinical studies within 4 weeks prior to informed consent
* Female subjects who are pregnant, possibly pregnant, or nursing, or who plan to become pregnant during the trial period
* Subjects otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Chair — Otsuka Pharmaceutical Co., Ltd.
Locations (5):
- Japan (5):
  - Chube Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-41061: Dose-titration period Administration of OPC-41061 will be started at 7.5 mg/day and the dose was increased stepwise up to as high as 60 mg/day until the dose for intermittent administration is determined. (If the dose was not fixed, the subject received the next higher dose following a 6-day washout period.) Intermittent administration period Subjects received once-daily 4-day intermittent administration of OPC-41061 (days on which hemodialysis or hemodiafiltration was not performed).
Period: Overall Study
Arm/Group | OPC-41061
Started | 23
Completed | 16
Not Completed | 7
Not completed — Lack of Efficacy | 5
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | OPC-41061
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Region of Enrollment [Number; unit: participants]
  Japan | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Urine Volume
Description: The daily urine volume at each timepoint and its change and the percent change from baseline will be summarized with descriptive statistics (number, mean, standard deviation [SD], minimum, median, maximum [same for following parameters]).
Time Frame: Baseline and Day 14 (Intermittent Administration Period)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | OPC-41061
Number analyzed (Participants) | 16
ml | 481.0 (427.1)

2. Secondary Outcome: Change From Baseline in Total Fluid Removal Per Week by Dialysis
Description: The total volume of fluid removed per week by dialysis at each timepoint and its change from baseline will be summarized with descriptive statistics.
Time Frame: Baseline (pretreatment observation period) and Intermittent Administration Period (Day 10 to Day 15)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | OPC-41061
Number analyzed (Participants) | 16
ml | -1425.0 (2139.7)

ADVERSE EVENTS:
Time Frame: From the start date of IMP administration to date of the final examination (up to Intermittent Administration Period Day15)
Arm/Group | OPC-41061
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 13/23
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 (N=23)
Thirst (General disorders) | 3
Malaise (General disorders) | 2
Injection site erosion (General disorders) | 1
Pyrexia (General disorders) | 1
Vessel puncture site pain (General disorders) | 1
Vessel puncture site pruritus (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 2
Periodontitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Blood urine present (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No